CLINICAL TRIAL: NCT07099144
Title: A Prospective, Open, Single-arm, Multi-center Phase IV Clinical Study of Inhaled Nitric Oxide Combined With Ventilatory Support for the Treatment of Neonatal (Gestational Age ≥34 Weeks) Hypoxic Respiratory Failure With Pulmonary Hypertension.
Brief Title: Inhaled Nitric Oxide for the Treatment of Neonatal Hypoxic Respiratory Failure With Pulmonary Hypertension
Acronym: INOFTTONHRFWPH
Status: Recruiting | Type: Observational
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: LeesPharm
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension; Hypoxic Respiratory Failure
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NO and NO2 concentration，Blood gas analysis，MetHb concentration，hematology panel (MetHb, RBC, WBC, PLT), biochemistry (AST, ALT, total bilirubin, direct bilirubin, BUN, creatinine), B-type natriuretic peptide (BNP), coagulation function (aPTT, PT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- inhaled nitric oxide combined with ventilatory support
  Interventions: Drug: Inhaled nitric oxide (NO)

INTERVENTIONS:
Drug: Inhaled nitric oxide (NO) — The starting dose of INOmax is 20 ppm, which is controlled by the INOmax DSIR Plus delivery system in the respiratory circuit during mechanical ventilation. The dose will be maintained at 20 ppm for 4 hours after the start of administration, then the dose can be weaned to 5 ppm provided that the arterial oxygenation is adequate, as determined by the investigator within 4-24 hours of therapy, and the therapy should be maintained at 5 ppm until the fraction of inspired oxygen (FiO2) < 0.60.
  The treatment will be maintained until the potential hypoxia is resolved, or the investigator determines that the neonate no longer needs to use this drug. The maintenance treatment time is usually less than 4 days (96 hours). If the oxygenation level has not improved significantly after 4 days of maintenance treatment, the suitability of the treatment plan should be reassessed.

SUMMARY:
This is a prospective, open-label, single-arm, multicenter Phase IV clinical study to evaluate the safety of INOmax for the treatment of hypoxic respiratory failure with pulmonary hypertension in newborns (≥ 34 weeks gestational age). To evaluate the safety of INOmax combined with ventilatory support in the treatment of neonatal (≥ 34 weeks gestational age) hypoxic respiratory failure with pulmonary hypertension.

DETAILED DESCRIPTION:
The study treatment will be administered in ventilated newborn infants expected to require support > 24 hours, after respiratory support has been optimized. This includes optimizing tidal volume/pressures and lung recruitment (surfactant, high frequency ventilation, and positive end expiratory pressure).

The administration of the study drug will be supervised by a physician investigator experienced in neonatal intensive care and used in clinics where neonatal artificial ventilation as well as rescue and resuscitation are available.

The starting dose of INOmax is 20 ppm, which is controlled by the INOmax DSIR Plus delivery system in the respiratory circuit during mechanical ventilation. The dose will be maintained at 20 ppm for 4 hours after the start of administration, then the dose can be weaned to 5 ppm provided that the arterial oxygenation is adequate, as determined by the investigator within 4-24 hours of therapy, and the therapy should be maintained at 5 ppm until the fraction of inspired oxygen (FiO2) < 0.60.

The treatment will be maintained until the potential hypoxia is resolved, or the investigator determines that the neonate no longer needs to use this drug. The maintenance treatment time is usually less than 4 days (96 hours). If the oxygenation level has not improved significantly after 4 days of maintenance treatment, the suitability of the treatment plan should be reassessed. If it is necessary to continue using this drug after evaluation by the investigator, the maximum administration time should not exceed 14 days.

Doses greater than 20 ppm are not allowed. Monitoring

1. Measure methemoglobin within 4-8 hours after initiation of treatment with INOmax and periodically throughout treatment.
2. Prior to INOmax treatment, appropriate procedures must be followed to purify the nitrogen dioxide (NO2) system so that the NO2 concentration should always be less than 0.5 ppm and maintained as low as possible, if NO2 is greater than 0.5 ppm, the delivery system will be assessed for failure, the NO2 analyzer will be recalibrated, and the dose and/or FiO2 will be reduced appropriately.
3. Monitor for inspired NO2 during INOmax administration.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates ≥ 34 weeks gestation age.
2. Hypoxic respiratory failure requiring more than 24 hours of ventilatory support.
3. Clinical or echocardiographic evidence of pulmonary hypertension (systolic pulmonary arterial pressure [sPAP] > 35 mm Hg or > 2/3 systemic blood pressure [SBP] or there is a right-to-left shunt at the atrium or arterial ductus).
4. Age less than 7 days at the time of treatment initiation with study drug.
5. The neonatal guardian agrees to participate in the study and signs an informed consent form (ICF).

Exclusion Criteria:

1. Neonates dependent on right-to-left shunting of blood.
2. Neonates whose mother has been treated with anticoagulant therapies during pregnancy.
3. Echocardiography confirmed left-to-right shunt or left ventricular dysfunction.
4. ECMO is urgently needed, or neonate has received ECMO.
5. Patient is at risk of imminent death (death expected within 24 hours).
6. Life-threatening abnormality (cranial, cardiac, thoracic).
7. Chromosomal abnormality.
8. Congenital diaphragmatic hernia
9. Congenital heart defect (other than patent ductus arteriosus or small atrial septal defect).
10. Neonate has been resuscitated requiring chest compressions within 6 hours of study treatment start.
11. Significant bleeding diathesis such as grade IV intraventricular hemorrhage or periventricular leukomalacia, pulmonary hemorrhage, uncontrolled bleeding or hemodynamic failure.
12. Disseminated intravascular coagulopathy.
13. Active seizures while receiving anticonvulsants.
14. Experienced prolong asphyxia with evidence of severe acidosis (pH<7.25)
15. Receiving nitric oxide donor agents such as prilocaine, sodium nitroprusside, nitroglycerin, and sulfonamides.
16. Other subjects determined by the investigator to be unsuitable for inclusion.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 120 neonates (gestational age ≥ 34 weeks) hypoxic respiratory failure with pulmonary hypertension.
  The study treatment will be administered in ventilated newborn infants expected to require support > 24 hours, after respiratory support has been optimized. This includes optimizing tidal volume/pressures and lung recruitment (surfactant, high frequency ventilation, and positive end expiratory pressure).
  The administration of the study drug will be supervised by a physician investigator experienced in neonatal intensive care and used in clinics where neonatal artificial ventilation as well as rescue and resuscitation are available.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of inhaled nitric oxide combined with ventilatory support in the treatment of neonatal (≥ 34 weeks gestational age) hypoxic respiratory failure with pulmonary hypertension. | Adverse events that occured during the study, not more than 14 days. Blood routine, blood biochemistry, blood gas analysis, chest X-ray and echocardiography will be performed at the screening and through study completion, not more than 14 days.
  Incidence and severity of all treatment emergent adverse events (TEAEs). Incidence of drug-related serious AEs (SAEs). Incidence of AEs of special interest (AESI).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children'S Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No